CLINICAL TRIAL: NCT03663062
Title: ObeSity Related Colorectal Adenoma Risk
Acronym: OSCAR
Status: Completed | Type: Observational
Sponsor: South Tyneside and Sunderland NHS Foundation Trust (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other); City Hospitals Sunderland NHS Foundation Trust (Other); North Tees and Hartlepool NHS Foundation Trust (Other); South Tees Hospitals NHS Foundation Trust (Other); Kettering General Hospital NHS Foundation Trust (Other); Royal Bolton Hospital NHS Foundation Trust (Other); Gloucestershire Hospitals NHS Foundation Trust (Other); University Hospitals of Morecambe Bay NHS Trust (Other); Mid Cheshire Hospitals NHS Foundation Trust (Other Government); Lancashire Teaching Hospitals NHS Foundation Trust (Other); Blackpool Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: OSCAR
Record Dates: First submitted 2017-12-15; First posted 2018-09-10 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2018-09

CONDITIONS: Colorectal Adenoma; Colorectal Neoplasm; Colorectal Cancer; Obesity; Metabolic Syndrome; Non-Alcoholic Fatty Liver Disease; Liver Fibrosis
Keywords: colorectal adenoma; colorectal cancer; Obesity; Non-Alcoholic Fatty Liver Disease; Metabolic syndrome; Liver Fibrosis
MeSH Terms: conditions — Colorectal Neoplasms; Obesity; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — Colonoscopy; Hematologic Tests; Blood Pressure; Medical History Taking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Colonoscopy — All patients would undergo colonoscopy as part of standard care. Patients recruited for this study would have their past medical history, family history, medication history, as well as waist circumference, BMI and blood pressure recorded. All patients would also have blood tests (described earlier) and a subset will undergo Fibroscan.
  Other Names: Blood tests; Fibroscan; BMI measurement; Waist circumference measurement; Blood pressure; Past medical history, family history, medication history

SUMMARY:
In the UK, around 1 in 16 men and 1 in 20 women will develop bowel cancer at some point in their lives. Most bowel cancers happen when a type of growth in the bowel called an adenoma eventually becomes cancerous. Cutting out adenomas reduces the risk of developing bowel cancer.

Certain people are more likely to have adenomas than others, for example people who are overweight. People who are overweight are also more likely to develop liver disease by laying too much fat down in the liver. Studies in Asia have shown that people with fatty liver disease are more likely to have adenomas and these are more commonly found in the part of the bowel (right colon) furthest from the bottom end.

Information on the link between obesity, fatty liver disease and adenomas is very limited, particularly in the Western population.

The investigators will assess the link between body weight, fatty liver and adenomas in the UK population. 1430 patients will be invited; some through the bowel cancer screening programme and some with symptoms such as low blood count, bleeding or changed bowel habit. These patients will already have been referred for a camera test looking into the bowel, called a colonoscopy. Information including height, weight and some health questions will be taken. Blood samples will be taken. The investigators will compare the number of patients with adenomas who have liver disease or who are overweight with those who don't. This information will be used to develop a scoring system to predict risk of adenomas. This will help the investigators to decide if undertaking colonoscopies in these patients will identify those at increased risk of bowel cancer.

DETAILED DESCRIPTION:
Bowel cancer, or colorectal cancer (CRC), is the second most common cancer affecting both men and women in England. The majority of CRCs develop from a pre-cancerous type of growth in the bowel called an adenoma. Detecting and removing these adenomas is important in reducing CRC risk. A study which undertook a once-off camera examination of the left hand side of the bowel (flexible sigmoidoscopy), removing any adenomas, demonstrated a reduction in CRC by 23% and reduced mortality by 31%.

Although a single cause for adenomas is not known, several factors can predispose patients to adenomas, including; age, gender, family history, cigarette smoking and excess body weight (EBW).

Obesity is becoming an increasing problem in the UK, with approximately a quarter of adults classed as obese in England. Patients who are obese are at higher risk of having adenomas. Studies have shown that patients with EBW are more likely to have fatty disease of the liver (non-alcoholic fatty liver disease, NAFLD) by laying down fat in the liver. Studies in Asia have shown that patients with NAFLD are more likely to have adenomas, and that these are more likely to be in the right side of the bowel which is furthest from the anus (right colon). Although these studies have shown a link between NAFLD and adenomas, they have all used invasive or expensive markers of fatty liver disease. No study has correlated the link between liver enzymes (blood tests) and adenomas or by using scoring systems to determine the presence or absence of significant fatty liver disease. Furthermore, no Western studies have confirmed the link between NAFLD and adenomas, meaning it is unclear whether this link is only present in the Asian population.

Approximately 400,000 colonoscopies (camera examinations of the large bowel) are performed each year within the NHS for the investigation of gastrointestinal symptoms, including: altered bowel habit, rectal bleeding and low blood count. When polyps are found, patients often have a follow-up surveillance colonoscopy to check that no new adenomas have formed. The timing and need for surveillance is based only on the number and size of adenomas found and does not take into account any risk factors which the patient may have.

The NHS Bowel Cancer Screening Programme (BCSP) invites all individuals aged 60-74 to undertake a stool sample test which looks for blood, called faecal occult blood testing (FOBt), every two years. Those who have a positive FOBt are then invited for a colonoscopy. This programme is purely based on age and is not targeted. Another arm of the BCSP was introduced in 2013, where all individuals aged 55 are invited for a flexible sigmoidoscopy and removal of adenomas. Anyone who is felt to be high risk according to the number or size of adenomas then undergoes a colonoscopy.

The BCSP has led to cancers being detected at an earlier stage, but is not protecting the population against cancers in the right side of the bowel.

In summary, although studies in Asian populations have suggested an association between NAFLD and colorectal adenomas, this has not been repeated in a Western population. It is important that the association is explored further in a Western population, in a simple, non-invasive manner. Assessing markers of NAFLD and a wider range of risk factors for adenomas will allow us to develop a tool to predict which patients are at increased risk of adenomas, called a risk model.

The OSCAR study is a multicentre observational study has been designed which will recruit 1430 participants from nine sites, eight in the North of England who are all members of the Northern Region Endoscopy Group (NREG) and one from Kettering General Hospital NHS Trust. NREG is an endoscopy research collaborative group with an excellent track record of delivering similar endoscopy based research studies to time and target. Participation will involve collecting information relating to obesity and fatty liver disease in patients already attending for colonoscopy in addition to collecting information about the number and size of any adenomas found.

All patients scheduled for colonoscopy will be provided with an invitation letter and patient information sheet in addition with the standard information about the colonoscopy procedure that the endoscopy unit provides. As colonoscopy requires a period of preparation prior to the test, patients will receive this information at least 24 hours before the procedure, allowing ample time to consider the study before attending the endoscopy department.

Taking part in this study will change very little about the patients' experience of the colonoscopy test itself. If the patient agrees to take part in this study, the information sheet will be reviewed with them by a research team member, an opportunity to ask questions given, and the consent form signed. Eligibility to take part in the study will be checked, and the patient will be weighed, have their height checked, waist circumference measured, body mass index (BMI) calculated and blood pressure checked. A research team member will undertake a health questionnaire which will include the following items:

1. Current and previous smoking history
2. Current and previous alcohol history
3. Current medications: including Aspirin, Statin, Insulin, non-steroidal anti-inflammatory drugs (NSAIDs), Diabetic medication, antibiotics and others
4. Family history of colorectal cancer
5. Family history of ischaemic heart disease in a first degree relative under the age of 60
6. History of liver disease
7. History of hypertension
8. History of diabetes- Type I, Type II
9. History of chronic kidney disease (Stage 4/5)
10. History of atrial fibrillation
11. History of rheumatoid arthritis
12. Personal history of anti-obesity surgery

These will be entered onto the case report form (CRF).

An intravenous cannula (a thin, plastic tube which is inserted into a vein in the arm) is then inserted as part of routine care before the colonoscopy procedure. Blood tests will be taken from this at the time of insertion to prevent the need for a separate blood test. These tests will include:

1. Bilirubin
2. Alanine aminotransferase (ALT)
3. Alkaline phosphatase (ALP)
4. Aspartate aminotransferase (AST)
5. Gamma-glutamyl transferase (GGT)
6. Full blood count (FBC)
7. HbA1c
8. Fasting blood glucose
9. Lipids: Cholesterol, HDL and Triglycerides
10. Albumin
11. Immunoglobulin A

Patients will also need to sign a separate consent form for the colonoscopy procedure itself as part of routine practice.

The patient will then enter the procedure room as per usual practice for their colonoscopy. During the procedure, the research team member will record data onto the CRF (procedural data, findings at colonoscopy etc). The colonoscopy report will be generated as per the usual practice in each unit.

A subset of patients will undergo Fibroscan, which is a non-invasive test to evaluate for liver fibrosis, to explore the association between the presence of colorectal adenoma/CRC and the presence of liver fibrosis.

After the procedure, the patient will enter the recovery ward and follow usual practice in the unit. Although participants will remain in the study for 14 days to allow data collection and to follow-up any abnormal results, participants will not require any further visits and the majority will not be contacted by the research team. If a new abnormality is found on checking blood samples, the patient will be contacted by a member of the research team and advised to make an appointment with their General Practitioner (GP).

Statistical analysis will be undertaken by Professor Steven Rushton, Professor of Biological Modelling at Newcastle University.

The primary outcome of this study is to develop a risk model which can be used to inform colorectal neoplasia screening and surveillance guidelines and to inform a future study targeting screening of higher risk individuals.

The secondary outcomes will support this model by identifying which demographics contribute to increased predisposition to colorectal neoplasia, namely smoking history, alcohol intake, and obesity (measured by BMI and waist circumference). The investigators also aim to assess whether the presence or degree of liver fibrosis, as measured by FIB4 score and Fibroscan affects the risk of colorectal neoplasia and by exploring the link between NAFLD, obesity and colorectal neoplasia in terms of adenoma burden, site and histological features. Lastly, the association between abnormal liver enzymes and colorectal neoplasia will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and over
2. Able to give informed consent
3. Indications:

   1. Patients with positive faecal occult blood test (FOBt) referred for index colonoscopy as part of Bowel Cancer Screening Programme
   2. Colonoscopy conversion from Bowelscope
   3. Index diagnostic colonoscopy due to new gastrointestinal symptoms (including but not restricted to diarrhoea, change in bowel habit, abdominal pain, PR bleeding, weight loss), iron deficiency anaemia, family history of CRC, abnormal findings on cross sectional imaging

Exclusion Criteria:

1. Absolute contraindication to colonoscopy
2. Unable to give informed consent
3. Known colorectal cancer
4. Known polyposis syndrome
5. Previous total/subtotal colectomy
6. Known colonic stricture which would prevent completion of colonoscopy
7. Attending for therapeutic procedure
8. Attending for assessment of a known lesion
9. Attending for assessment of known inflammatory bowel disease (IBD)
10. Attending for surveillance colonoscopy (polyp surveillance, post colorectal cancer surveillance, IBD surveillance)
11. Colonoscopy within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient referred for colonoscopy matching the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 1430 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Risk model of colorectal adenomas and CRC | 24 months from patient recruitment
  Risk prediction model

SECONDARY OUTCOMES:
The incidence of colorectal adenomas or CRC in patients with abnormal liver enzymes | 24 months from patient recruitment
  Number of patients with colorectal adenomas or CRC who have abnormal liver enzymes
The incidence colorectal adenomas or CRC in patients with obesity | 24 months from patient recruitment
  Number of patients with colorectal adenomas or CRC who are obese, as measured by BMI or waist circumference
The incidence colorectal adenomas or CRC in patients with abnormal FIB4 score | 24 months from patient recruitment
  Number of patients with colorectal adenomas or CRC who have abnormal FIB4 score
The incidence colorectal adenomas or CRC in patients with abnormal Fibroscan readings | 24 months from patient recruitment
  Number of patients with colorectal adenomas or CRC who have abnormal Fibroscan readings
The incidence of colorectal adenomas or CRC in patients who are smokers or who have high alcohol intake | 24 months from patient recruitment
  Number of patients with colorectal adenomas or CRC who are smokers or have high alcohol intake

CONTACTS AND LOCATIONS:
Overall Officials: Colin Rees, FRCP, Principal Investigator — South Tyneside and Sunderland NHS Foundation Trust
Locations (12):
- United Kingdom (12):
  - Royal Bolton Hospital, Bolton, Greater Manchaster
  - University Hospitals of Morecambe Bay NHS Foundation Trust, Lancaster, Lancashire
  - Mid Cheshire Hospitals NHS Foundation Trust, Crewe, Mid Cheshire
  - South Tyneside NHS Foundation Trust, South Shields, Tyne and Wear
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucester
  - Kettering General Hospitals NHS Foundation Trust, Kettering
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Newcastle Upon Tyne NHS Foundation Trust, Newcastle upon Tyne
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - North Tees and Hartlepool NHS Foundation Trust, Stockton-on-Tees
  - CIty Hospitals Sunderland NHS Foundation Trust, Sunderland

IPD SHARING:
Plan to Share IPD: No
There are no plans for this at present

DOCUMENTS (2):
  • Study Protocol (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT03663062/Prot_000.pdf
  • Informed Consent Form (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT03663062/ICF_001.pdf